CLINICAL TRIAL: NCT03986840
Title: Effectiveness of the Multicomponent Exercise Training in Frail Elderly
Brief Title: Multicomponent Exercise Training in Frail Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Carlos Romero Morales, Senior Lecturer, PhD, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIPI/
Record Dates: First submitted 2019-06-07; First posted 2019-06-14 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Frailty; Exercise Addiction
Keywords: Frailty; Exercise; Aging
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise program (Experimental): The exercise program was applied for 6 weeks. A total of 18 sessions were distributed in 3 weekly sessions. The participants performed a resistance exercises: leg press at an intensity of 40%-60% with 10 repetitions, 12 repetitions of steps with their bodyweight and a plantar flexion followed by a cardiovascular HIIT exercise walking on a treadmill.
  Interventions: Other: Exercise training
- Daily activities (Active Comparator): The patients who belongs to this group will continue to perform their daily routines.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — A multicomponent exercise program

SUMMARY:
The aim of the present study will be to assess the effectiveness of the multicomponent exercise training in frail for the physical function, frailty and performance.

All the individuals will be assessed two times.

DETAILED DESCRIPTION:
This will be a experimental, randomized controlled intervention study in frail. Subjects will be recruited at the Albertia Care Center, Madrid. The exercise training group will developed a concurrent training 3 days per week during 6 weeks. The control group will follow an usual care also for 6 weeks.

The main variables will be as follows:

* Ultrasound imaging measurements for the lower limb: core muscles, vastus medialis, rectus femoris, vastus intermedius, gastrocnemius, soleus. We will employed a General Electric (GE) Ultrasound device in B mode to assess the thickness of the muscles.
* Heart rate variability with a Suunto smart bell.
* Activities of daily living with the Bartel index.
* Force-velocity profile and muscle power.
* Frailty with the Linda´s frailty criteria.

The exercise program was applied for 6 weeks. A total of 18 sessions were distributed in 3 weekly sessions. The participants performed a resistance exercises: leg press at an intensity of 40%-60% with 10 repetitions, 12 repetitions of steps with their bodyweight and a plantar flexion followed by a cardiovascular high intensity interval training (HIIT) exercise walking on a treadmill.

One measurements will be taken (pre), the second (post) measurements will be performed at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 75 years or more,
* 2 or more points in the Short Physical Performance Battery (SPPB)
* Capability of walking (alone or assisted)

Exclusion Criteria:

* Severity cognitive alterations
* Severe disability on the Barthel score
* Surgeries in the previous 6 months
* Other any disorder that exclude for the exercise group.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
Thickness of the core and quadriceps muscles | Change from baseline muscle thickness at 6 weeks
  Thickness assessment by ultrasound imaging
Heart rate variability | Change from baseline heart rate variability at 6 weeks
  Heart rate variability by Suunto smart bell device
Daily life activities | Change from baseline daily life activities at 6 weeks
  Bartel index questionnaire
Muscle power | Change from baseline muscle power at 6 weeks
  Force-velocity profile for the lower limb muscle power
Frailty | Change from baseline frailty at 6 weeks
  Frailty with the Linda´s frailty criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sergio López, MsC, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Albertia Elderly Care Center, Madrid, Spain